CLINICAL TRIAL: NCT04736758
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study on the Safety and Efficacy of GP681 Tablets in the Treatment of Uncomplicated Acute Influenza
Brief Title: A Clinical Study on the Safety and Efficacy of GP681 Tablets in the Treatment of Uncomplicated Acute Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP681-202002
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GP681 tablet 40mg (Experimental): Patients in the GP681 tablet 40mg group is treated with GP681 tablet 40mg orally once with 240mL water.
  Interventions: Drug: GP681 tablet
- GP681 tablet 20mg (Experimental): Patients in the GP681 tablet 40mg group is treated with GP681 tablet 20mg orally once with 240mL water.
  Interventions: Drug: GP681 tablet
- Placebo group (Placebo Comparator): Patients in the Placebo group is treated with GP681 Simulant orally once with 240mL water.
  Interventions: Drug: GP681 Simulant

INTERVENTIONS:
Drug: GP681 tablet — influenza subjects is randomized 1:1:1 into GP681 tablet 40mg group,GP681 tablet 20mg group and Placebo group,with 72 patients in each group.subjects is given with GP681 tablet or GP681 Simulant only once to treat influenza.
  Arms: GP681 tablet 20mg; GP681 tablet 40mg
Drug: GP681 Simulant — influenza subjects is randomized 1:1:1 into GP681 tablet 40mg group,GP681 tablet 20mg group and Placebo group,with 72 patients in each group.subjects is given with GP681 tablet or GP681 Simulant only once to treat influenza.
  Arms: Placebo group

SUMMARY:
Analyse the time of flu symptom relief in adults with uncomplicated acute influenza,to evaluate the antiviral effects of high and low doses of GP681 tablets, and explore the optimal dose for phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Positive Influenza rapid antigen test;
* Fever (axillary temperature ≥37.3℃) or the axillary temperature ≥37.3℃ after taking the medicine for more than 4 hours;
* At least one systemic symptom and respiratory symptom related to a moderate or above influenza virus infection:

  1. Systemic symptoms: headache, fever or chills, muscle or joint aches, fatigue;
  2. Respiratory system symptoms: cough, sore throat, nasal congestion.
* Time of disease symptoms ≤48h

Exclusion Criteria:

* Diagnosed as severe influenza patient ;
* Known history of dysphagia or any gastrointestinal disease that affects drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, stomach After subtotal resection, etc.);
* Have used anti-influenza virus drugs (oseltamivir, zanamivir, peramivir, favipiravir, abidol, baloxavir dipivoxil, amantadine, or diamond) within 2 weeks before screening Ethylamine, etc.);
* Acute respiratory infections, otitis media, sinusitis or other infectious diseases such as bronchitis, pneumonia, tuberculosis, etc. occurred within 2 weeks before screening, and are in the acute stage;
* Patients who also suffer from bacterial or viral infections and need systemic antibacterial or antiviral therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
time to alleviation of influenza symptoms | Day 15
  Defined as the time from the start of treatment until the patient's body temperature returns to normal and all 7 flu symptoms (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, fatigue) have alleviated (scoring 0 or 1 point) .

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, phd, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Wang H, Liu D, Ding Y, Zhang M, Xiao Z, Jiang X, Wu Y, Zhang W, Sun S, Chen X, Zhang W, Tang Y, Jiang M, Yang G, Jia W, Wang X, Tong J, Suo L, Yu Y, Yan X, Li Z, Li X, Cao B. Efficacy and safety of single-dose suraxavir marboxil tablet in the treatment of acute uncomplicated influenza in adults: a multi-centre, randomized, double-blind, placebo-controlled phase 2 clinical trial. Clin Microbiol Infect. 2025 May;31(5):861-868. doi: 10.1016/j.cmi.2025.01.025. Epub 2025 Jan 25. PMID 39870350